CLINICAL TRIAL: NCT02451046
Title: Predictive Ability of Alpha-GST to Detect Graft Primary Dysfunction After Liver Transplantation
Brief Title: Usefulness of Alpha-GST in Liver Transplantation
Acronym: GST-LT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beaujon Hospital (Other)
Responsible Party: Principal Investigator, Paugam-Burtz, Professor, Beaujon Hospital
Other Study IDs: 2015-A00839-40
Record Dates: First submitted 2015-05-19; First posted 2015-05-21 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Evidence of Liver Transplantation
Keywords: Liver transplantation; Primary dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary objective of this study was to evaluate the ability of plasma alpha-GST measurements in liver donor (at the time of organ removal) to predict primary dysfunction in liver recipient. The secondary objective was to study the relationship between alpha-GST levels in the plasma of the liver transplant recipient and early graft function recovery.

DETAILED DESCRIPTION:
Graft primary dysfunction (PDF) after liver transplantation is enhanced by the increasing use of extended-criteria allografts. This complication is burdened with high mortality and morbidity rates among liver transplant recipients. Alpha-GST is a short-life hepatocyte enzyme that may be an interesting biomarker for liver injury. A recently developped ELISA technique may allow fast and easy measurement of alpha-GST plasma concentration (Fastpack IP α-GST Immunoassay, Qualigen Inc., Carlsbad, CA). This study aims to evaluate the ability of plasma alpha-GST measurements in liver donor to predict PDF in liver recipient. Methods: Observational study conducted in one center (Beaujon hospital, APHP, Clichy, France). Measurements of plasma levels of alpha-GST using Fastpack IP α-GST Immunoassay (Qualigen Inc., Carlsbad, CA) at the time of organ removal in liver donor and daily from day 0 to day 7 after liver transplantation in recipients.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* undergoing liver transplantation at Beaujon hospital (APHP, Clichy, France )

Exclusion Criteria:

* age >70 years and <18 years

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing liver transplantation at Beaujon hospital (APHP, Clichy, France)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-03; Primary Completion 2015-10 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Primary dysfunction (PDF) of liver graft | First week
  To evaluate the ability of plasma alpha-GST measurements in liver donor (at the time of organ removal) to PDF in liver recipient.

SECONDARY OUTCOMES:
Early graft function recovery. | First week
  To study the relationship between alpha-GST levels in the plasma of the liver transplant recipient and early graft function recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Paugam-Burtz, MD-PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Réanimation hépato-digestive, Clichy, France